CLINICAL TRIAL: NCT00012324
Title: A Phase III Randomized Controlled Study Comparing the Survival of Patients With Unresectable Hepatocellular Carcinoma (HCC) Treated With THYMITAQ to Patients Treated With Doxorubicin
Brief Title: Nolatrexed Dihydrochloride Compared With Doxorubicin in Treating Patients With Recurrent or Unresectable Liver Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eximias Pharmaceutical (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: ZARIX-ZX101-301; CDR0000068506 (Registry Identifier: PDQ (Physician Data Query)); AG-337-301
Record Dates: First submitted 2001-03-03; First posted 2003-01-27 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2005-10

CONDITIONS: Liver Cancer
Keywords: localized unresectable adult primary liver cancer; advanced adult primary liver cancer; recurrent adult primary liver cancer; adult primary hepatocellular carcinoma
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Doxorubicin; nolatrexed

INTERVENTIONS:
Drug: doxorubicin hydrochloride
Drug: nolatrexed dihydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known which chemotherapy regimen is more effective for liver cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of two different chemotherapy regimens in treating patients who have recurrent or unresectable liver cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival in patients with unresectable or recurrent hepatocellular carcinoma treated with nolatrexed dihydrochloride vs doxorubicin.
* Compare time to progression, time to treatment failure, and response rates in patients treated with these regimens.
* Compare the probability of survival at 3, 6, 9, and 12 months in patients treated with these regimens.
* Compare the safety and clinical benefit of these regimens in these patients.
* Compare the response rates and survival of patients who have received prior therapy or no prior therapy after treatment with these two regimens.
* Compare the rates of conversion from unresectable to resectable lesions in patients treated with these regimens.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to CLIP score (0-1 vs 2-3) and Karnofsky performance status (60-70% vs 80-100%). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive nolatrexed dihydrochloride IV continuously on days 1-5.
* Arm II: Patients receive doxorubicin IV on day 1. Treatment continues in both arms every 3 weeks in the absence of unacceptable toxicity or disease progression.

Patients are followed every 2 months for survival.

PROJECTED ACCRUAL: Approximately 446 patients (223 per treatment arm) will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven or presumptive diagnosis of hepatocellular carcinoma

  * Presumptive diagnosis based on rising alpha-fetoprotein (AFP) levels over 2 assessments, CT scan or MRI of liver, spiral CT scan of portal/splenic vein, and biopsy evidence of cirrhosis
  * Unresectable or recurrent disease after prior surgical resection or embolization therapy
* Fibrolamellar histology allowed if considered surgically unresectable based on tumor size, extrahepatic involvement, or multiple lobe involvement
* CLIP (Cancer of the Liver Italian Program) score less than 4
* Concurrent assignment to a transplantation list allowed

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,200/mm^3
* Platelet count at least 80,000/mm^3

Hepatic:

* Bilirubin no greater than 3.0 mg/dL (except for known Gilbert's Syndrome)
* AST no greater than 5 times upper limit of normal (ULN)
* PT no greater than 1.5 times ULN

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No uncontrolled hypertension within the past 3 months
* No unstable angina, symptomatic congestive heart failure, or myocardial infarction within the past 3 months
* No uncontrolled cardiac arrhythmia

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active bacterial infections
* HIV negative
* No AIDS
* No other primary malignancy except carcinoma in situ of the cervix or urinary bladder or non-melanoma skin cancer
* No mental incapacitation or psychiatric illness that would preclude study participation
* No other severe disease that would preclude study participation
* Candidate for placement of a central venous access device

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior biologic therapy allowed
* No concurrent biologic therapy

Chemotherapy:

* No prior IV doxorubicin except intraarterial administration in locoregional therapy

Endocrine therapy:

* Prior endocrine therapy allowed
* No concurrent endocrine therapy

Radiotherapy:

* Prior radiotherapy allowed
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics
* Surgery allowed if previously unresectable lesions become resectable
* Recovered from any prior surgery
* No concurrent liver transplantation

Other:

* No other concurrent investigational or marketed anticancer drugs
* No other concurrent therapy for hepatocellular carcinoma
* No concurrent terfenadine, astemizole, or cisapride that may not be interrupted during nolatrexed dihydrochloride administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-09; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Time to progression
Time to treatment failure
Response rate (complete response, partial response, stable disease)
Survival probabilities at 3, 6, 9, and 12 months
Safety
Response to treatment in patients with and without prior therapy

CONTACTS AND LOCATIONS:
Overall Officials: Gregory R. Suplick, Study Chair — Eximias Pharmaceutical
Locations (42):
- United States (38):
  - Arizona Clinical Research Center, Incorporated, Tucson, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Scripps Cancer Center at Scripps Clinic, La Jolla, California
  - David and Donna Long Center for Cancer Treatment at Sharp Grossmont Hospital, La Mesa, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - California Pacific Medical Center - Pacific Campus, San Francisco, California
  - Olive View - UCLA Medical Center Foundation, Sylmar, California
  - California Hematology/Oncology Medical Group, Torrance, California
  - Helen F. Graham Cancer Center, Newark, Delaware
  - Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Florida Cancer Institute - Bayonet Point, Hudson, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Oncology-Hematology Group of South Florida, P.A., Miami, Florida
  - Ocala Research Institute, Incorporated, Ocala, Florida
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - University of Illinois at Chicago Cancer Center, Chicago, Illinois
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Louisiana Oncology Associates - Lafayette, Lafayette, Louisiana
  - Stanley S. Scott Cancer Center at Louisiana State University Medical Center - New Orleans, New Orleans, Louisiana
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Saint Louis University Cancer Center, St Louis, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Cancer Centers of the Carolinas - Eastside, Greenville, South Carolina
  - Medical City Dallas Hospital, Dallas, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
- Canada (3):
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Ottawa Hospital Regional Cancer Centre - General Campus, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
- Fundacion de Investagacion De Diego, Santurce, Puerto Rico

REFERENCES:
- [Result] Gish RG, Porta C, Lazar L, Ruff P, Feld R, Croitoru A, Feun L, Jeziorski K, Leighton J, Gallo J, Kennealey GT. Phase III randomized controlled trial comparing the survival of patients with unresectable hepatocellular carcinoma treated with nolatrexed or doxorubicin. J Clin Oncol. 2007 Jul 20;25(21):3069-75. doi: 10.1200/JCO.2006.08.4046. PMID 17634485